CLINICAL TRIAL: NCT03530462
Title: The Usage of Neuropsychological Tests and Multi-mode Magnetic Resonance Imaging in Patients With Autoimmune Encephalitis for Cognitive Neural Mechanism
Brief Title: To Explore Cognitive Neural Mechanism of Autoimmune Encephalitis by Using Neuropsychological Tests and Multi-modal MRI
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: multi-mode MRIs- encephalitis
Record Dates: First submitted 2018-03-18; First posted 2018-05-21 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-02

CONDITIONS: Cognitive Impairment; Autoimmune Encephalitis
Keywords: episodic memory; executive control; fMRI
MeSH Terms: conditions — Cognitive Dysfunction; Autoimmune Diseases of the Nervous System | interventions — Rituximab; Cyclophosphamide; Steroids; Methylprednisolone; Immunoglobulins, Intravenous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patient with first-line and second-line: patients who received intravenous second-line immunotherapy (steroids, intravenous immunoglobulin, plasmapheresis),in addition to first-line immunotherapy (rituximab, cyclophosphamide)
  Interventions: Drug: rituximab; Drug: cyclophosphamide; Drug: Steroids; Drug: Intravenous immunoglobulin
- patients with first-line only: patients who received first-line immunotherapy (steroids, intravenous immunoglobulin, plasmapheresis)only
  Interventions: Drug: Steroids; Drug: Intravenous immunoglobulin
- healthy control: healthy individuals without a history of psychiatric or neurologic disease

INTERVENTIONS:
Drug: rituximab — 375 mg/m2 weekly for 4 weeks
  Other Names: rituximab injection
  Groups: patient with first-line and second-line
Drug: cyclophosphamide — 750 mg/m2 monthly for 4-6 cycles depending on the response
  Other Names: cyclophosphamide injection
  Groups: patient with first-line and second-line
Drug: Steroids — 500-1000 mg of methylprednisolone daily for 3 days, then tapered doses
  Other Names: methylprednisolone
  Groups: patient with first-line and second-line; patients with first-line only
Drug: Intravenous immunoglobulin — intravenous immunoglobulin (IVIG) with or without plasmapheresis
  Other Names: IVIG
  Groups: patient with first-line and second-line; patients with first-line only

SUMMARY:
Most of patients with autoimmune encephalitis are left with permanent cognitive deficits of varying severity. The patients' life and career would be affected definitely by cognitive deficits. Recently, more and more clinical physician have begun to focus on cognitive impairment of patients with autoimmune encephalitis. Generally, the outcome was measured by the modified Rankin Scale (mRS). However, the mRS are commonly used to evaluate the degree of disability or dependence in the daily activities of the patients suffering from a stroke and cognition function were minimally evaluated in this scale. It is crucial to adopt detailed cognition tools to study the long-term cognitive outcomes and as an indicator of overall curative effect judgment in autoimmune encephalitis.

Currently, only early immunotherapy is uniformly and consistently considered to produce favorable cognitive outcomes. However, studies concerning the association of second-line immunotherapy with cognitive outcomes have been scarce and have shown conflicting results regarding autoimmune encephalitis.

Hence, the goal of this study was to explore cognitive neural mechanism of autoimmune encephalitis by using neuropsychological tests and multi-mode MRIs.

DETAILED DESCRIPTION:
The goal of this study was to explore cognitive neural mechanism of different types of autoimmune encephalitis by using neuropsychological tests and multi-mode MRIs. Neuropsychological tests involves the assessments of different cognitive domains. And multi-mode MRIs contains resting-fMRI, DTI and task-related fMRI.

ELIGIBILITY:
Inclusion Criteria: Diagnosis was established in all patients based on characteristic clinical presentation and detection of immunoglobulin G (IgG) antibodies.

-

Exclusion Criteria:

1. age >60 years or <16 years
2. notable lesions, such as tumors, scars, or vascular malformations, on brain MRI
3. a history of other neuropsychiatric disorders. -

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: patients with autoimmune encephalitis and healthy control
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
brain functional connectivity changes | a minimum of 6 months following initial discharge from hospital
  The study uses multi-model fMRI to measure changes of functional connectivity across regions during recovery

SECONDARY OUTCOMES:
verbal episodic memory | a minimum of 6 months following initial discharge from hospital
  Chinese auditory verbal learning test (CAVLT)
non-verbal episodic memory | a minimum of 6 months following initial discharge from hospital
  Aggie Figures Learning Test (AFLT)
working memory | a minimum of 6 months following initial discharge from hospital
  working memory test
emotion-anxiety | a minimum of 6 months following initial discharge from hospital
  self-rating anxiety scale (SAS),the *total* range (20-80 scores), anxiety state (the total score is equal or above 41)
emotion-depression | a minimum of 6 months following initial discharge from hospital
  self-rating depression scale (SDS), the *total* range (20-80 scores), depression state (the total score is equal or above 41)
executive control | a minimum of 6 months following initial discharge from hospital
  Stroop test
information processing speed | a minimum of 6 months following initial discharge from hospital
  symbol-digit modalities test (SDMT)
visual-spatial ability | a minimum of 6 months following initial discharge from hospital
  block design test
semantic fluency test | a minimum of 6 months following initial discharge from hospital
  vegetable and fruit, animal

CONTACTS AND LOCATIONS:
Overall Officials: Benyan Luo, Ph.D, Principal Investigator — The First Affiliated Hospital, Zhejiang University
Locations (1):
- The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No